CLINICAL TRIAL: NCT04114123
Title: The Development of Reward Response to Food in Infancy
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Julie Lumeng, Thomas P Borders Family Research Professor of Child Behavior and Development, Professor of Pediatrics, Associate Dean for Research, Medical School, Professor of Nutritional Sciences, University of Michigan
Other Study IDs: HUM00164906
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Eating Behavior
Keywords: Reward-driven Eating; Infant; Maternal
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Longitudinal: The researchers will be evaluating baseline indicators of wanting salience and liking between 2 and 6 month olds, with the goal of following up with these families at 24 months and beyond by reviewing the dyads' medical charts. The researchers will also examine direct and indirect associations between reward-driven eating, and maternal and infant characteristics and infant weight-for-length.
- Cross-sectional: The researchers will as the mother to answer questionnaires and participate in up to two video taped behavioral protocols when the infant is 6 months old.

SUMMARY:
In this study the researchers want to learn more about reward-driven eating behavior in children ages 2 to 18 months. The researchers hope to use this knowledge to help inform obesity prevention programs.

DETAILED DESCRIPTION:
The study will comprise two arms and each arm has a different time perspective. The longitudinal arm is prospective in nature and the cross-sectional arm has a cross-sectional time perspective. The video observation is completed at a single time point (although standardized by inclusion criteria).

ELIGIBILITY:
For the Longitudinal Arm:

Inclusion Criteria

* Baby is alive
* Baby is 6 to 16 weeks old at time of enrollment
* Baby and mother receive care at Michigan Medicine, and specifically:

  * Baby was born at Michigan medicine
  * Baby has had a 2 month well child check
  * Mother received prenatal care at Michigan Medicine
  * Mother has a linked patient profile to baby's profile
  * Baby has a length and weight measurement on record
* Mother is English speaking

Exclusion Criteria

* Baby is a foster child
* Baby was still in hospital 4 days after birth
* Baby has severe perinatal or neonatal medical problems
* Baby has severe developmental delays
* Multiple births

For the Cross Sectional:

Inclusion Criteria

* Enrolled in longitudinal arm of study
* Eligible to complete all three protocols (Two Oatmeal and Reaching) as per protocol screeners
* Baby is alive
* Baby is 5 to 7 months old at the time of enrollment
* Mother is biological mother
* Mother is legal guardian
* Mother is English speaking

Exclusion Criteria

* Baby had severe perinatal or neonatal medical problems
* Baby currently has severe medical problems
* Baby has severe developmental delays
* Mom had severe complications during pregnancy
* Multiple Births
* Food allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The researchers will enroll infants and their mothers (age limit given is for minimum age for mothers) from the community and from sites allowed and approved by the IRB like pediatric clinics and childcare centers. They will be recruiting participants living within a 50 mile radius around Ann Arbor, MI.
Sampling Method: Non-Probability Sample
Enrollment: 1166 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Association of trajectory membership and body mass index z-score (BMIz) | Time Frame: 24 months
  Trajectory membership could be "wanting", "salience", or "liking"

OTHER OUTCOMES:
Association of reward-driven eating component wanting with maternal and infant characteristics | Up to 18 months
Association of reward-driven eating component salience with maternal and infant characteristics | Up to 18 months
Association of reward-driven eating component liking with maternal and infant characteristics | Up to 18 months
Association of maternal and infant characteristics and weight-for-length z-score (WLZ) | 2 months through 24 months
Association of infant reward-driven eating and weight-for-length z-score (WLZ) | 2 months through 24 months
Association of infant reward-driven eating and infant diet | Up to 18 months
Association of infant reward-driven eating and infant weight-for-length z-score (WLZ) | 6 months through 24 months
Association of infant diet and infant weight-for-length z-score (WLZ) | 6 months through 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lumeng, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The research will generate demographic, anthropometric, dietary, behavioral questionnaire, and coded behavioral data. (Note the researchers will not make video data available.) The data will be stored as Statistical Package for the Social Sciences (SPSS) or Statistical Analysis System (SAS) files. Meta data will also be included in the selected repositories.The meta data will include the data dictionaries, which describe the generation of all variables, as well as the protocol manuals describing the behavioral protocols used to generate the variables.
Time Frame: Data submitted to Deep Blue Data will be reviewed after 10 years to determine if a dataset should be retained and will be subject to further, periodic, reviews thereafter.
Access Criteria: All data in the Deep Blue Data repository are available to anyone for download without restriction.